CLINICAL TRIAL: NCT00073125
Title: A Phase II Randomized Study Evaluating the Safety and Efficacy of ABT-510 in Subjects With Advanced Renal Cell Carcinoma
Brief Title: Safety and Efficacy of ABT-510 in Subjects With Advanced Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M02-428; NCT00080704 (obsolete NCT alias)
Record Dates: First submitted 2003-11-17; First posted 2003-11-18 (Estimated); Last update posted 2007-08-15 (Estimated); Status verified 2007-08

CONDITIONS: Carcinoma, Renal Cell
Keywords: Advanced histologically documented renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ABT-510/Thrombospondin-1 mimetic

SUMMARY:
The primary objective of this study is to assess the safety and efficacy of ABT-510 in subjects with advanced renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for study participation if all of the following criteria are met:

* The subject is at least 18 years of age.
* The subject has advanced histologically documented renal cell carcinoma. Advanced disease is defined as locally recurrent disease or metastatic disease that is not amendable to curative resection.
* The subject has not received prior therapy (anti-tumor radiotherapy, immunotherapy, chemotherapy, or investigational therapy) for metastatic renal cell carcinoma other than excision of primary tumor where appropriate. Local radiation for supportive reasons will be allowed; however, not within 28 days from Study Day 1.
* The subject has an Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-1
* The subject is able to self-administer or has a caregiver who can reliably administer subcutaneous injections.
* The subject must have adequate bone marrow, renal, and hepatic function as follows:

  * Bone Marrow: White blood cell count (WBC) ≥ 3,000/mm3 (3.0 X 109/L); Platelets ≥ 100,000/mm3 (100 X 109/L); Hemoglobin ≥ 9.0 g/dL (1.4 mmol/L)
  * Renal function: serum creatinine ≤ 2.0 mg/dL (0.81 mmol/L)
  * Hepatic function: AST and ALT ≤ 1.5 X ULN unless liver metastases are present, then AST and ALT ≤ 5.0 X ULN; LDH ≤ 1.5 X ULN; bilirubin ≤ 1.5 mg/dL (0.026 mmol/L) Corrected calculated calcium ≤ 10 mg/dL (2.5 mmol/L) Calculation = total calcium - 0.707 (albumin -3.4)Albumin ≥ 3.0 g/dL (0.45 mmol/L)
* The subject must not be pregnant or lactating and all subjects (male and female) must use a contraceptive method deemed acceptable by the investigator while in the study and for up to two months following completion of therapy.
* The subject has voluntarily signed and dated an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved consent prior to any study specific procedures.

Exclusion Criteria:

A subject will be ineligible for study participation if any of the following criteria are met:

* The subject has a history of or currently exhibits Central Nervous System (CNS) metastasis. Brain MRI within 28 days of enrollment is required to confirm absence of CNS metastases.
* The subject is receiving therapeutic anticoagulation therapy. Low dose anticoagulation (e.g., low dose Coumadin) for catheter prophylaxis will be permitted; PT/PTT must be within normal limits.
* The subject has a history of or currently exhibits clinically significant cancer related events of bleeding (e.g., hemoptysis). The subject has a recent history of (within 4 weeks of Study Day 1) or currently exhibits other clinically significant signs of bleeding.
* The subject exhibits evidence of clinically significant uncontrolled conditions(s) and/or is considered by the investigator to be unable to tolerate the proposed treatment or procedures.
* The subject has history of other previous malignancies within 5 years, with the exception of: Adequately treated in situ carcinoma of the cervix uteri or Basal or squamous cell carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2003-05

PRIMARY OUTCOMES:
Progression free survival | One year

SECONDARY OUTCOMES:
Response rate | One year
Overall survival | One year
Performance status | One year

CONTACTS AND LOCATIONS:
Overall Officials: Rod Humerickhouse, MD, Study Director — Abbott
Locations (17):
- United States (16):
  - Virginia G. Piper Cancer Center, Scottsdale, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - UCLA School of Medicine, Los Angeles, California
  - Clinical Trials and Research Associates, Montebello, California
  - The Center for Hematology-Oncology, Boca Raton, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Central indiana Cancer Center, Indianapolis, Indiana
  - Kansas City Cancer Centers Southwest, Overland Park, Kansas
  - University of Michigan, Ann Arbor, Michigan
  - Kansas City Oncology and Hematology Group, Kansas City, Missouri
  - Albany Regional Cancer Center, Albany, New York
  - Raleigh Hematology Oncology Clinic, Cary, North Carolina
  - US Oncology, P.A., Dallas, Texas
  - Texas Cancer Center, Fort Worth, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
- Academic Hospital Groningen, Groningen, Netherlands